CLINICAL TRIAL: NCT06531837
Title: Electroencephalographic Characteristics of Chronic Pain in Patients With Spinal Cord Injury: an Exploratory, Interventional, Non-randomized Controlled Study
Brief Title: Electroencephalographic Characteristics of Chronic Pain in Patients With Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: zz20240512
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain
Keywords: Multichannel electroencephalogram; patients with spinal cord injury; Esketamine; Remifentanil; Flurbiprofen; Spinal cord stimulation
MeSH Terms: conditions — Chronic Pain | interventions — Remifentanil; Flurbiprofen; Injections, Intravenous; Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients without pain (Sham Comparator)
  Interventions: Other: No intervention
- Patients with chronic pain treated with esketamine (Experimental)
  Interventions: Drug: Esketamine(Continuous infusion); Device: Spinal Cord Stimulation
- Patients with chronic pain treated with remifentanil (Experimental)
  Interventions: Drug: Remifentanil (Target-Controlled Infusion); Device: Spinal Cord Stimulation
- Patients with chronic pain treated with flurbiprofen (Experimental)
  Interventions: Drug: Flurbiprofen (Single intravenous injection); Device: Spinal Cord Stimulation

INTERVENTIONS:
Drug: Esketamine(Continuous infusion) — Continuous intravenous infusion of esketamine at a dose of 0.2 mg/(kg · h). Collect resting-state EEG data and NRS scores 40 minutes after administration.
  Arms: Patients with chronic pain treated with esketamine
Drug: Remifentanil (Target-Controlled Infusion) — The plasma drug concentrations of remifentanil were set at 0.5 ng/ml, 1 ng/ml, and 1.5 ng/ml. After each plasma drug concentration reached a steady state, the NRS scores were assessed, and resting-state EEG was recorded for at least 5 minutes.
  Arms: Patients with chronic pain treated with remifentanil
Drug: Flurbiprofen (Single intravenous injection) — Single intravenous injection of Flurbiprofen at a dose of 100 mg. Collect resting-state EEG data and NRS scores 10 minutes after administration.
  Arms: Patients with chronic pain treated with flurbiprofen
Device: Spinal Cord Stimulation — Collect resting-state EEG data and NRS scores with the spinal cord stimulator both turned off and on.
  Arms: Patients with chronic pain treated with esketamine; Patients with chronic pain treated with flurbiprofen; Patients with chronic pain treated with remifentanil
Other: No intervention — Collect resting-state EEG data and NRS scores.
  Arms: Patients without pain

SUMMARY:
The diagnosis of chronic pain currently lacks objective and quantifiable biomarkers. This study aims to observe the EEG characteristics of patients with chronic pain following spinal cord injury and subsequently administer analgesic interventions with remifentanil, esketamine, flurbiprofen, and spinal cord stimulation. The correlation between EEG features and pain intensity will be examined. The research aims to advance the objectification of chronic pain diagnosis and treatment.

ELIGIBILITY:
Spinal Cord Injury Patients With Chronic Pain

Inclusion Criteria:

* Age 18 - 65 years old;
* American Society of Anesthesiologists (ASA) I-III;
* Dextromanual;
* Chronic Pain following Spinal Cord Injury;
* Spinal cord electrical stimulator implantation under general anesthesia;
* Signed informed consent.

Exclusion Criteria:

* People with mental and behavioral disorders.
* Previous history of craniocerebral disease;
* History of drug and alcohol abuse;
* Patients with aphasia or inability to cooperate with the pain assessments;
* Previous adverse reaction to esketamine, opioids or NSAIDs;
* Known sever insufficiency of vitals(such as heart failure/renal dysfunction/hepatic failure);
* Patients with myasthenia gravis, bronchial asthma, or a predisposition to respiratory depression;
* Bleeding tendency;
* BMI ≥ 35 kg/m²;
* Pregnancy or lactation.

Spinal Cord Injury Patients Without Pain

Inclusion Criteria:

* Age 18 - 65 years old;
* American Society of Anesthesiologists (ASA) I-III;
* Dextromanual;
* Spinal Cord Injury Patients Without Pain;
* Spinal cord electrical stimulator implantation under general anesthesia;
* Signed informed consent.

Exclusion Criteria:

* People with mental and behavioral disorders.
* Previous history of craniocerebral disease;
* History of drug and alcohol abuse;
* Patients with aphasia or inability to cooperate with the pain assessments;
* Previous adverse reaction to esketamine, opioids or NSAIDs;
* Known sever insufficiency of vitals(such as heart failure/renal dysfunction/hepatic failure);
* Patients with myasthenia gravis, bronchial asthma, or a predisposition to respiratory depression;
* Bleeding tendency;
* BMI ≥ 35 kg/m²;
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
EEG Spectral Characteristics | During the trial(up to 3 hours for each subject).
  EEG power spectrum characteristics of chronic pain in patients with spinal cord injury under esketamine, remifentanil, flurbiprofen administration and spinal cord stimulation, including the δ, θ, α, β, and γ frequency bands.
  administration, including the δ, θ, α, β, and γ frequency bands.

SECONDARY OUTCOMES:
Numeric Rating Scale(NRS) | During the trial(through study completion, 7 days)
  Numerical Rating Scale Assessment Pre- and Post-Analgesic Treatment. The NRS ranges from 0 to 10, with 0-3 indicating mild pain, 4-6 indicating moderate pain, and 7-10 indicating severe pain.
Generalized Anxiety Disorder(GAD-7) | During the trial(through study completion, 7 days)
  The GAD-7 scale ranges from 0 to 21 points, with a higher score indicating a higher level of anxiety.
Patient Health Questionnaire-9(PHQ-9) | During the trial(through study completion, 7 days)
  The PHQ-9 scale ranges from 0 to 27 points, with a higher score indicating a higher level of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph D, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China